CLINICAL TRIAL: NCT06979778
Title: A Randomized Controlled Trial to Assess the Efficacy of the "Syd" App on Improving Quality of Life and Mental Health Among University Students in the Kingdom of Saudi Arabia
Brief Title: Testing the Efficacy of the "Syd" App on Improving Quality of Life and Mental Health Among University Students in the Kingdom of Saudi Arabia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iamYiam Limited (Industry)
Collaborators: Alfaisal University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250512
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Quality of Life (QOL); Anxiety; Stress; Affect (Mental Function)
Keywords: syd; QoL; See Yourself Differently; Quality of Life; mHealth; App; RCT
MeSH Terms: conditions — Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- syd app (Experimental): The 'syd' application is designed as an AI-powered "Life Quality Mentor" with the primary aim of enhancing users' quality of life. The app focuses on positive habit development, personalised feedback, and continuous support. It offers personalised guidance across various domains, including Physical health, Emotional health, Brain power, Self-awareness, Purpose, Career, Financial health, Social life and Environment. It utilizes an advanced AI platform and offers features like personalised recommendations, supportive interaction with an AI mentor, habit tracking tools, and integration with wearable technology.
  The intervention arm will have full access to the 'syd' app and be able to interact with it for the 3 months duration of the trial
  Interventions: Device: See Yourself Differently (syd) mobile app
- Wait list control (No Intervention): The wait list control arm will not receive access to the 'syd' app for the 3 months' duration of the trial, but will be given full lifetime access thereafter.

INTERVENTIONS:
Device: See Yourself Differently (syd) mobile app — The 'syd' mobile app is designed as an AI-powered "Life Quality Mentor" with the primary aim of enhancing users' quality of life. The app focuses on positive habit development, personalised feedback, and continuous support. It offers personalised guidance across various domains, including Physical health, Emotional health, Brain power, Self-awareness, Purpose, Career, Financial health, Social life and Environment. It utilizes an advanced AI platform and offers features like personalised recommendations, supportive interaction with an AI mentor, habit tracking tools, and integration with wearable technology.
  Other Names: syd; See Yourself Differently
  Arms: syd app

SUMMARY:
The goal of this clinical trial is to learn if using the "See Yourself Differently" (syd) app can help improve quality of life and mental health for university students in Saudi Arabia. The study also aims to see if the app can help lower anxiety and stress, and increase positive feelings while decreasing negative feelings.

The main questions it aims to answer are:

1. Does the "syd" app improve the quality of life for university students?
2. Does the "syd" app help lower anxiety and stress in university students
3. Does the "syd" app help increase positive feelings and decrease negative feelings in university students?

Researchers will compare students who use the "syd" app to see if it works.

Participants will:

1. Use the "syd" app for 3 months.
2. Complete surveys about their quality of life, anxiety, stress, and feelings.

DETAILED DESCRIPTION:
This clinical trial outlines a prospective, parallel-group, single-blind randomised controlled trial to be conducted at Alfaisal University in the Kingdom of Saudi Arabia. The study will enrol 600 university students and staff members and will run for a 3-month intervention period.

The intervention focuses on the 'syd' mobile application, an AI-powered "Life Quality Mentor" designed to enhance users' quality of life. The app aims to support positive habit development by providing personalised feedback and continuous support. Key features include personalised guidance across various domains such as nutrition, sleep performance, stress management (including guided meditations and journaling), and financial well-being. The 'syd' app utilizes an advanced Artificial Intelligence (AI) platform, offering an AI conversational agent for motivational coaching, habit tracking tools, and integration with wearable technology.

Participants will be randomly allocated to either an experimental group, which will use the 'syd' app, or a control group. Those in the experimental group will be instructed to use the 'syd' app for the 3-month duration of the study.

Data will be collected at multiple time points: at baseline (prior to intervention), monthly during the 3-month intervention period, and at a final follow-up post-intervention. The primary data collection methods will involve validated research instruments (WHOQOL-BREF, PANAS-X, GAD-7, PSS) administered via Typeform surveys. Additionally, in-app data will be collected to monitor app usage, specifically the frequency and duration of engagement. Socio-demographic information will also be gathered.

Survey data will be stored securely within Typeform, and in-app data will be stored within the 'syd' application's database, hosted securely on Amazon Web Services (AWS). All data storage will comply with Alfaisal University's data security policies. To protect participant privacy, data will be anonymised or de-identified where possible, and access will be restricted to authorised research team members. Data will be encrypted during storage and transmission.

For data analysis, linear mixed-effects modelling will be employed, incorporating random intercepts for participants and fixed effects for time, group, and the time x group interaction. The analysis will adhere to intention-to-treat principles. Should missing data occur, multiple imputation will be considered if feasible. Data from Typeform surveys will be exported and cleaned, in-app data will be extracted and processed, and data from these different sources will be merged for comprehensive analysis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Enrolled as a full-time medical student at the Alfaisal university.
* Owning a smartphone (iOS or Android) compatible with the "syd" app.
* Willing to provide informed consent and comply with study procedures

Exclusion Criteria:

* Known severe psychiatric or cognitive conditions that impede app usage
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life Domain Scores | From enrolment to the end of treatment at 3 months
  Quality of Life (QoL) as measured through the WHOQOL-BREF instrument. The WHOQOL-BREF is a 26-item questionnaire which uses a scoring system that assesses quality of life across four domains: physical health, psychological health, social relationships, and environmental health. Each item is scored on a 5-point scale (1-5) and transformed to a 0-100 scale. Domain scores are calculated by summing relevant item scores and transforming them to a 0-100 scale. Higher scores indicate better quality of life in a specific domain.

SECONDARY OUTCOMES:
Change in Anxiety Score | From enrolment to the end of treatment at 3 months
  Change in Anxiety scores as measured through the General Anxiety Disorder-7 (GAD-7) questionnaire. The GAD-7 scoring system uses a simple system to assess anxiety levels. Each of the seven questions on the GAD-7 questionnaire is scored from 0 to 3, with 0 representing "not at all" and 3 representing "nearly every day." The total score is calculated by adding up the scores for all seven questions, resulting in a total score ranging from 0 to 21. Score interpretation: 0-4: Minimal to no anxiety; 5-9: Mild anxiety; 10-14: Moderate anxiety; 15 or higher: Severe anxiety.
Change in Perceived Stress Score | From enrolment to the end of treatment at 3 months
  Change in Perceived Stress Score as measured through the Perceived Stress Scale (PSS) questionnaire. The PSS scores are determined by summing individual item responses and interpreting the total score. Higher scores indicate a higher level of perceived stress. The total score can range from 0 to 56, with higher scores reflecting higher levels of stress.
Change in Positive and Negative Affect Scores | From enrolment to the end of treatment at 3 months
  Change in Positive and Negative Affect Scores as measured through the Positive and Negative Affect Schedule - Expanded Version (PANAS-X) questionnaire. The PANAS-X is composed of 60 items (emotions) on a 5-point scale (1 to 5) where participants can indicating how much they feel each emotion. A total positive and negative affect score is calculated by summing the responses for the respective sets of items. Higher scores on the positive affect scale indicate greater positive affect, while lower scores on the negative affect scale indicate less negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abu-Zaid, MD, Principal Investigator — Alfaisal University
Locations (1):
- Alfaisal University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No